CLINICAL TRIAL: NCT04518527
Title: Evaluation of Short-term and Residual Effects of Kinesio Taping in Chronic Lateral Epicondylitis: A Randomized, Double-blinded, Controlled Trial
Brief Title: Efficiency of Kinesio Taping in Chronic Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Balevi Batur (Other)
Responsible Party: Sponsor-Investigator, Elif Balevi Batur, Assistant Prof, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziU
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2017-02

CONDITIONS: Tendinopathy, Elbow
Keywords: Kinesio taping; lateral epicondylitis; residual effect
MeSH Terms: conditions — Elbow Tendinopathy; Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- true taping+ exercise (Active Comparator): The true taping method was applied to the first group according to the method determined by Kase. According to this method, a 2-inch (5 cm) wide beige-colored Kinesio tape (Kinesio® Tex Gold FP) was measured from the second-third metacarpal base to the lateral epicondyle while the elbow was extended and the wrist was in the neutral position and the tape was applied in the shape of a 'Y'. In a position where the wrist-ankle extensors were most tense (wrist-ankle extension - forearm pronation), the anchor point of the tape was applied to the insertion of the muscle without creating any tension. Then, the tape was applied to the medial and lateral edges of the wrist extensors by applying a 15-25% tension towards the origin of the muscle. Both ends of the Y-shaped tape were terminated without tension on the lateral epicondyle.
  Interventions: Device: Tape
- sham taping+exercise (Placebo Comparator): In the placebo group, the 10 cm I-shaped tape was placed 5 cm inferior to the lateral epicondyle using the same Kinesio tape in the study group. It was applied transversely, starting from the painless side of the midline on the forearm extensor face directing towards the lateral side of the forearm without a tension.
  Interventions: Device: Tape

INTERVENTIONS:
Device: Tape — The tape is an elastic cotton strip with an acrylic adhesive that is used with the intent of treating pain and disability

SUMMARY:
Lateral epicondylitis is a degenerative tendinosis of the extensor carpi radialis brevis muscle and is the most common work/sports-related chronic musculoskeletal problem affecting the elbow. This randomized, double-blinded, controlled study aimed to evaluate the short term and residual effectiveness of the Kinesio taping method on pain, grip force, quality of life, and functionality.

DETAILED DESCRIPTION:
Fifty patients diagnosed with chronic unilateral lateral epicondylitis with a symptom duration of at least 12 weeks. The study group received a true inhibitor Kinesio taping while the control group received sham taping for the first four weeks. In both groups, progressive stretching and strengthening exercises were given as a home program for 6 weeks. Patients were assessed with the numerical rating scale (NRS), Cyriax resistive muscle test evaluation, maximal grip strength, PRTEE (Patient- Rated Tennis Elbow Evaluation), and SF-36 (Short Form-36) by the first assessor who was blinded to taping types.

ELIGIBILITY:
Inclusion Criteria:

* Having pain on or near the lateral epicondyle and increases with pain at least one of the following provocations tests for lateral epicondylitis -resisted wrist extension (Cozen's test), resisted elbow supination (Mill's test) and 3rd finger extension (Maudley's test),
* Unilateral elbow pain at least 12 weeks,
* Not received injection therapy to the elbow in the last six weeks,
* Not received a physical therapy program in the last three months,
* Presence of normal elbow radiographic findings,
* Normal elbow joint range of motion,
* Having no neurological deficits

Exclusion Criteria:

* Patients with degenerative joint disease,
* Radial tunnel syndrome,
* Cervical nerve root compression,
* Pain reflected from the neck, shoulders,
* Wrist, radiohumeral joint osteochondritis dissecans,
* Tendon rupture,
* Osteoporosis, Infection,
* Malignancy,
* Inflammatory disease,
* Pregnant women

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
numerical rating scale | 1 year
  The numerical rating scale (NRS) was used to evaluate the pain level of the patients included in the study. It is a one-dimensional scale consisting of 11 items that measure pain intensity in adults and is a segmented - intermittent numerical version of the visual analogue scale (VAS).

SECONDARY OUTCOMES:
resisted muscle test evaluation | 1 year
  According to the Cyriax method, each joint tested was kept in the mid- range of motion, without allowing movement. Resistance was applied to the forearm distal to avoid muscle involvement other than that tested in pronation and supination, thus the wrist was prevented to be involved. Subsequently, the patients were asked to apply a maximum force for at least three seconds. Resisted wrist extension, third finger extension, elbow supination, and pronation were evaluated.
Maximal Isometric Handgrip Strength | 1 year
  The maximal isometric handgrip strength was measured in pounds using the Jamar hand dynamometer (Baseline® Hand Dynamometer - HiRes™ Gauge - ER™ 300 lbCapacity). Measurement was performed in two different positions, elbow at extension and 90° flexion. In the first position, the patient was in the sitting position, shoulder abducted to 0° and in neutral rotation, elbow position was at 90° flexion, the forearm was in neutral rotation and wrist was in the neutral position. In the second position, while the patient was standing, shoulder abducted to 0° and in neutral rotation, the elbow was in full extension, forearm and wrist were in the neutral position. The patient was asked to squeeze the dynamometer with full force for three seconds every 30 seconds. This procedure was repeated three times and the mean measurement values were obtained
The Patient-rated Tennis Elbow Evaluation(PRTEE) | 1 year
  The Patient-rated Tennis Elbow Evaluation (PRTEE) is a questionnaire with subscales related to pain and function, which is used to evaluate upper extremity functionality. It is specially prepared for patients with lateral epicondylitis.Scoring ranges from 0 (no pain/disability) to 100 (worst possible pain and disability). The total score can be 100 points maximum and low scores refer to better functionality.Turkish validity and reliability was proven by Altan et al.
36-Item Short-Form Health Survey (SF-36) | 1 year
  The SF-36 is valid and reliable for patients with chronic musculoskeletal disorders. The items include eight different domains that indicate physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation, and mental health. The score of each domain ranges from 0 (worst quality of life) to 100 (the best quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: IŞIL S YENİCE BALEVİ, Principal Investigator — Gazi University; BELGİN KARAOĞLAN, Study Director — Gazi University; NAGİHAN ACET, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).